CLINICAL TRIAL: NCT00049608
Title: A Phase I Study Of The Effect Of Mistletoe Extract, A Complementary Medicine Botanical, On Pharmacokinetics, Pharmacodynamics And Safety Of Gemcitabine In Patients With Advanced Solid Tumors
Brief Title: Gemcitabine Combined With Mistletoe in Treating Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal investigator [PI] has left institution.
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258130; NCCAM-02-AT-260; NCI-02-AT-0260; NCT00044161 (obsolete NCT alias)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2007-04

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Pancreatic Cancer
Keywords: male breast cancer; recurrent breast cancer; recurrent colon cancer; recurrent non-small cell lung cancer; recurrent pancreatic cancer; recurrent rectal cancer; stage III colon cancer; stage III pancreatic cancer; stage III rectal cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; stage IV colon cancer; stage IV non-small cell lung cancer; stage IV rectal cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Breast Neoplasms, Male; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung; Rectal Neoplasms | interventions — Gemcitabine

INTERVENTIONS:
Dietary Supplement: mistletoe extract
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, use different ways to stop tumor cells from dividing so they stop growing or die. Mistletoe may slow the growth of tumor cells and may be an effective treatment for solid tumors.

PURPOSE: Phase I trial to study the effectiveness of combining gemcitabine with mistletoe in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of gemcitabine and mistletoe in patients with advanced solid tumors.
* Determine the toxic effects of this regimen in these patients.
* Determine the pharmacokinetic effects of gemcitabine with and without mistletoe in these patients.
* Determine tumor response in patients treated with this regimen.
* Determine the time to neutrophil count recovery in patients treated with this regimen.

OUTLINE: This is an open-label, dose-escalation study.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and mistletoe subcutaneously daily starting on day 8 of course 1. Treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

Patients receive escalating doses of gemcitabine and mistletoe in 2 stages.

* Stage I: Cohorts of 3-6 patients receive escalating doses of mistletoe in combination with a constant dose of gemcitabine until the maximum tolerated dose (MTD) of mistletoe is determined.
* Stage II: Cohorts of 3-6 patients receive escalating doses of gemcitabine in combination with the MTD of mistletoe as determined in stage I until the MTD of gemcitabine is determined.

In both stages, the MTD is defined as the dose preceding that at which 2 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 45-51 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic, recurrent, or unresectable locally advanced solid tumor, including one of the following:

  * Breast or colorectal cancer that has failed first-line chemotherapy
  * Non-small cell lung cancer
  * Pancreatic Cancer
* No CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* No clinically significant hepatic dysfunction

Renal

* Creatinine no greater than 2.5 mg/dL
* No clinically significant renal dysfunction

Other

* Not pregnant or nursing
* Negative pregnancy test
* HIV negative
* No clinically significant unrelated illness (e.g., serious infection or organ dysfunction) that would preclude study tolerance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior mistletoe

Chemotherapy

* See Disease Characteristics
* No prior gemcitabine
* More than 30 days since prior chemotherapy and recovered

Endocrine therapy

* More than 30 days since prior glucocorticosteroid therapy

Radiotherapy

* Recovered from prior radiotherapy

Surgery

* Recovered from prior surgery

Other

* At least 30 days since prior investigational agents
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2002-07; Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Mansky, MD, Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

REFERENCES:
- [Result] Mansky PJ, Wallerstedt DB, Sannes TS, Stagl J, Johnson LL, Blackman MR, Grem JL, Swain SM, Monahan BP. NCCAM/NCI Phase 1 Study of Mistletoe Extract and Gemcitabine in Patients with Advanced Solid Tumors. Evid Based Complement Alternat Med. 2013;2013:964592. doi: 10.1155/2013/964592. Epub 2013 Oct 27. PMID 24285980